CLINICAL TRIAL: NCT02726737
Title: Effect of Sodium Bicarbonate Buccal Infiltration on the Success of Inferior Alveolar Nerve Block in the Mandibular First Molar With Symptomatic Irreversible Pulpitis: a Prospective, Randomized Double-blind Study
Brief Title: Effect of Sodium Bicarbonate Buccal Infiltration on the Success of Inferior Alveolar Nerve Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Masoud Saatchi (Other)
Responsible Party: Sponsor-Investigator, Masoud Saatchi, Professor of Endodontics, School of Dentistry, Isfahan University of Medical Sciences, Isfahan University of Medical Sciences
Organization: Isfahan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 941456
Record Dates: First submitted 2016-03-30; First posted 2016-04-04 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-02

CONDITIONS: Local Anesthesia
Keywords: inferior alveolar nerve block; irreversible pulpitis; local anesthesia; sodium bicarbonate
MeSH Terms: interventions — Sodium Bicarbonate; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sodium bicarbonate (Experimental): 0.7 mL of 8.4% sodium bicarbonate & 0.3 mL of 2% lidocaine with 1:100,000 epinephrine
  Interventions: Drug: sodium bicarbonate; Drug: Lidocaine
- Non-sodium bicarbonate (Active Comparator): Sterile distilled water & 0.3 mL of 2% lidocaine with 1:100,000 epinephrine
  Interventions: Drug: Lidocaine; Drug: sterile distilled water

INTERVENTIONS:
Drug: sodium bicarbonate
  Arms: sodium bicarbonate
Drug: Lidocaine
Drug: sterile distilled water
  Arms: Non-sodium bicarbonate

SUMMARY:
The purpose of this prospective, randomized, double blind study was to evaluate the effect of a buccal infiltration of sodium bicarbonate on the anesthetic success of the inferior alveolar nerve block (IANB) in patients with mandibular first molar experiencing symptomatic

DETAILED DESCRIPTION:
Several studies have been done by adding Sodium Bicarbonate to local anesthesia in dentistry based on the theory that the amount of local anesthetic in the free-base un-ionized form will decrease to provide greater lipid penetration of the nerve and this could be cause of the failure of local anesthesia injected into the inflamed tissue with low PH and conflicting results were obtained. But, there are no study that evaluate effect of increasing PH in periradicular tissue on hindrance of resistance channels with supplementary infiltration injection of Sodium Bicarbonate

ELIGIBILITY:
Inclusion Criteria:

* vital mandibular molar tooth
* diagnosis of symptomatic irreversible pulpitis

Exclusion Criteria:

* younger than 18 years old
* history of significant medical conditions
* allergies to local anesthetics or sulfites
* pregnancy
* taking any medications that might influence anesthetic assessment
* active sites of pathosis in area of injection
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
success rate of IANB in the mandibular first molar with symptomatic irreversible pulpitis | Baseline

SECONDARY OUTCOMES:
Heft-Parker visual analog scale recording of pain | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Saatchi, Study Chair — Isfahan University of Medical Sciences
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No